CLINICAL TRIAL: NCT04762602
Title: A Multicenter, Open-Label, Phase I Study Evaluating the Safety and Tolerability of HMPL-306 in Subjects With Advanced or Metastatic Solid Tumors With IDH Mutations
Brief Title: A Study of HMPL-306 in Advanced Solid Tumors With IDH Mutations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated based on strategic evaluation of the clinical development of HMPL-306 with no safety concerns
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-306-GLOB2
Record Dates: First submitted 2021-02-06; First posted 2021-02-21 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Isocitrate Dehydrogenase Gene Mutation
Keywords: Cholangiocarcinoma; Skeletal chondrosarcoma; Glioma; IDH Mutation
MeSH Terms: conditions — Cholangiocarcinoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Dose Escalation Cohorts (Experimental): Patients from each cohort will be administered HMPL-306 orally QD
  Interventions: Drug: HMPL-306
- Part 2 Dose Expansion Cohorts (Experimental): Patients from each cohort will be administered HMPL-306 orally QD at the recommended phase 2 dose
  Interventions: Drug: HMPL-306

INTERVENTIONS:
Drug: HMPL-306 — Administered orally QD in a 28-day continuous dosing treatment cycle

SUMMARY:
An open label single-arm clinical trial to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of HMPL-306 in advanced or metastatic solid tumors with IDH mutation.

DETAILED DESCRIPTION:
HMPL-306 is a dual IDH1/2 inhibitor

This is a phase 1, open-label, multicenter study to evaluate the safety and tolerability of HMPL-306 administered orally in the treatment of subjects with advanced or metastatic solid tumors with IDH mutation. The study consists of 2 parts: Part 1 (dose escalation) and Part 2 (dose expansion). The dose escalation part will determine the MTD/RP2D. The dose expansion part will administer the MTD/RP2D to mIDH-positive solid tumor malignancies including, but not limited to, cholangiocarcinoma, skeletal chondrosarcoma, low-grade glioma, perioperative low-grade glioma

ELIGIBILITY:
Key Inclusion Criteria:

Subjects are eligible for enrollment into this study if they meet any of the following criteria (NOTE: This is not an exhaustive list):

* Subjects aged ≥18 years.
* ECOG performance status 0 or 1
* Subjects must have a documented IDH mutation per immunohistochemistry (IHC), polymerase chain reaction (PCR), or next generation sequencing (NGS) testing of tumor tissue.
* Subjects must have histologically or cytologically documented, advanced or metastatic solid malignancy of any type that has recurred or progressed on available standard treatment and for which no curative therapy exists.

Key Exclusion Criteria:

Subjects are not eligible for enrollment into this study if they meet any of the following criteria (NOTE: This is not an exhaustive list):

* Subjects who received an investigational agent <14 days prior to their first day of study drug administration
* Subjects who are pregnant or breastfeeding
* Subjects with an active severe infection, some treated infections and with an expected or with an unexplained fever >38.3°C during screening visits or on their first day of study drug administration.
* Subjects with some current or prior heart conditions
* Subjects taking medications that are known to prolong the QT interval may not be eligible
* Subjects with immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation
* Some subjects with some current or prior gastrointestinal or liver diseases
* Subjects with inadequate organ function as defined by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Subjects with Dose Limiting Toxicities (DLTs) | Up to 28 days after first dose of study drug
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 and is at least possibly related to study drug.
Part 1 and Part 2: Frequency and severity of AEs | From the first dose of the study drug to 37 days after the last dose of study drug

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From first dose of study drug to the time of progressive disease, assessed up to 36 months
  ORR is defined as the proportion of subjects with confirmed best overall tumor response of Complete Response (CR) or Partial Response (PR).
Clinical Benefit Rate (CBR) | From first dose of study drug to the time of progressive disease, assessed up to 36 months
  CBR is the proportion of subjects with stable disease (SD), confirmed PR or confirmed CR (CR+PR+SD).
Duration of response (DoR) | From first dose of study drug to the time of disease relapse or death, whichever comes first, assessed up to 36 months
  DoR defined as the time from the date of the first CR or PR to the first date of progressive disease (PD) or death from any cause.
Progression-free Survival (PFS) | From first dose of study drug to the time of progressive disease or death due to any causes, whichever comes first, assessed up to 36 months
  PFS is defined as time from first dose date of study drug to date of progression or date of death from any cause, whichever occurred first.
Maximum serum drug concentration | PK weeks at screening through safety follow-up, assessed up to 36 months
  Blood samples will be obtained from all patients for determination of the maximum serum concentration of HMPL-306
Time to maximum concentration | PK weeks at screening through safety follow-up, assessed up to 36 months
  Blood samples will be obtained from all patients for determination time to maximum concentration of HMPL-306
Area under the concentration-time curve (AUC) | PK weeks at screening through safety follow-up, assessed up to 36 months
  Blood samples will be obtained from all patients for determination of the AUC of HMPL-306

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhang, Study Director — Hutchison Medipharma Limited
Locations (11):
- United States (8):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer, Pittsburgh, Pennsylvania
  - Houston Methodist, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Spain (3):
  - Hospital de la Santa creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid